CLINICAL TRIAL: NCT05257590
Title: A Phase 2, Open-Label Study of CVM-1118 in Combination With Nivolumab in Subjects With Unresectable Advanced Hepatocellular Carcinoma
Brief Title: CVM-1118 in Combination With Nivolumab for Unresectable Advanced Hepatocellular Carcinoma
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: TaiRx, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CVM-008
Record Dates: First submitted 2022-02-08; First posted 2022-02-25 (Actual); Last update posted 2025-12-17 (Actual); Status verified 2025-12

CONDITIONS: Hepatocellular Carcinoma; Advanced Cancer
Keywords: Oncology; Hepatocellular Carcinoma (HCC); Nivolumab; Hepatoma
MeSH Terms: conditions — Carcinoma, Hepatocellular; Neoplasms | interventions — Nivolumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Nivolumab + CVM-1118 (Experimental): 1 Cycle = 28 days
  Nivolumab, 240 mg, IV, Q2 weeks with an option for 480 mg, IV, Q4 weeks starting from Cycle 3 if judged to be reasonable by the investigator based on the safety and tolerability.
  CVM-1118, 200 mg, PO, BID with an option to increase the starting dose to 300 mg, PO, BID for the subsequent subjects following assessment of safety data from the initial 10 subjects. Escalation of the starting dose will be dependent on the absence of Dose Limiting Toxicity in at least 7 of the initial 10 subjects treated at 200 mg, PO, BID.
  Individual subjects receiving a starting dose of 200 mg, PO, BID and who tolerate the initial 2 cycles with no more than Grade 2 related toxicity, will have the option of increasing their dose of CVM-1118 to 300 mg, PO, BID (600 mg total daily dose) starting with cycle 3
  Tolerable dose of Nivolumab and CVM-1118 will be administered continuously for a 28-day cycle until progressive disease, unacceptable toxicity, or consent withdrawal.
  Interventions: Drug: Nivolumab Injection [Opdivo]; Drug: CVM-1118

INTERVENTIONS:
Drug: Nivolumab Injection [Opdivo] — Nivolumab will be administered at 240 mg, IV, Q2 weeks with an option for 480 mg, IV, Q4 weeks starting with Cycle 3 if judged to be reasonable by the investigator based on the safety and tolerability.
  Other Names: Nivolumab
Drug: CVM-1118 — CVM-1118 will be administered 200 mg, PO, BID with an option to increase the starting dose to 300 mg, PO, BID for the subsequent subjects following assessment of safety data from the initial 10 subjects.
  Other Names: TRX-818

SUMMARY:
CVM-1118 is a new small molecule chemical entity being developed as a potential anti-cancer therapeutic by TaiRx, Inc. CVM-1118 is a potent anti-cancer agent in numerous human cancer cell lines. The safety of administrating CVM-1118 on human has been evaluated from the phase 1 study. The objective of the phase 2 study is to further investigate the efficacy of CVM-1118 with nivolumab for subjects with unresectable advanced hepatoma.

DETAILED DESCRIPTION:
Nivolumab, a human IgG4 kappa monoclonal antibody acts as a checkpoint inhibitor, blocking the interaction between PD-1 and its ligands (PD-L1 and PD-L2 ) and therefore preventing the activation of T cells from attacking the cancer. Nivolumab is currently approved for several cancer types.

To meet the medical need, TaiRx, Inc. develops a new small molecule drug, CVM-1118 can promote apoptosis and delay proliferation. Moreover, CVM-1118 targets the formation of vasculogenic mimicry (VM). VM has been associated with tumor metastasis and poor clinical outcomes. VM is reported to be particularly active in tumor under hypoxia state when patients are treated with the potent vascular endothelial growth factor (VEGF) inhibitor like sorafenib or bevacizumab. Hence, the ability of inhibiting the VM network makes CVM-1118 a potential good combination drug with Nivolumab in advanced diseases such as hepatoma where Nivolumab alone has shown activity.

The safety profile of CVM-1118 dosing has been established in the phase 1 study. The analysis of metabolism pathways further showed that the potential drug-drug interactions of CVM-1118 and Nivolumab are very low.

Based on the mechanism of actions and the safety analysis of nivolumab and CVM-1118, the design of phase 2 trial with the combination therapy might have great potential for the patients with unresectable advanced HCC.

ELIGIBILITY:
Inclusion Criteria:

* Age 18+ (20+ for subjects in Taiwan)
* Diagnosis of hepatocellular carcinoma

  * Pathologically or cytologically-confirmed or clinically diagnosed in accordance with American Association for the Study of Liver Diseases (AASLD) criteria (i.e., radiologic imaging with cross-sectional multiphasic contrast CT or MRI showing a ≥ 1 cm liver lesion)
* Subjects with advanced-stage, unresectable hepatocellular carcinoma that is not appropriate for potentially curable therapy who have progressed from, been intolerant of prior systemic anti-cancer therapies (e.g., sorafenib, lenvatinib, atezolizumab in combination with bevacizumab).
* Barcelona Clinic Liver Cancer (BCLC) stage B not appropriate for or with disease progression after local regional therapy, or BCLC stage C
* Child-Pugh liver function class A
* Measurable disease (per mRECIST)
* ECOG performance status of 0 to 1
* Adequate laboratory parameters including:

  * AST and ALT ≤ 3.0 x ULN (≤ 5.0 x ULN if due to liver involvement)
  * Total serum bilirubin ≤ 2.0 x ULN (≤ 3.0 x ULN for subjects with documented Gilbert's syndrome)
  * ANC ≥1500/µL
  * Platelets ≥ 90,000/µL
  * HGB ≥ 9.0 g/dL
  * Serum creatinine clearance of ≥ 50 mL/min based on Cockcroft-Gault formula
  * Serum albumin ≥ 2.8 gm/dL
  * INR ≤ 2.3
  * PT/aPTT ≤ 1.2 x ULN
* QTcF ≤ 480 msec
* Subjects are eligible to enroll if they have HBV-, or HCV-HCC, defined as follows:

  * Chronic HBV infection as evidenced by detectable HBV DNA or HBsAg. Subjects with chronic HBV infection must be on antiviral therapy and have HBV DNA <500 IU/mL. If not on an antiviral therapy at screening, then subjects must be willing to start the antiviral therapy at the time of consent.
  * Active or resolved HCV infection as evidenced by detectable HCV RNA or antibody.

Exclusion Criteria:

* HCC with portal vein invasion at the main portal branch (Vp4)
* Known history of esophageal varices or gastrointestinal bleeding within the past 3 months
* Prior immunotherapy for hepatoma
* ≤ 7 days from prior limited field palliative irradiation therapy and C1D1
* ≤ 28 days from prior irradiation therapy and C1D1
* ≤ 14 days (or 5 half-lives) from prior systemic anticancer therapy and C1D1
* ≤ 28 days from local regional therapy (e.g., trans-arterial embolization, radiofrequency ablation) and C1D1
* Presence of other active cancer(s) likely to require treatment in the next two (2) years or likely to impact the assessment of any study endpoints
* Active bacterial or fungal infection(s) requiring systemic therapy within 7 days prior to C1D1
* Known CNS metastases
* Known history of HIV infection
* Females who are currently pregnant or breast-feeding
* Known gastrointestinal disease that may significantly alter the absorption of oral medications
* Psychiatric illness or social situation that would interfere with compliance with study requirements
* History of clinically significant cardiovascular abnormalities

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 95 (Estimated)
Dates: Start 2022-05-23 (Actual); Primary Completion 2026-03-31 (Estimated); Study Completion 2026-03-31 (Estimated)

PRIMARY OUTCOMES:
Objective Response Rate (ORR)_mRECIST | 24 weeks after the last subject starts CVM-1118
  Assessment by modified RECIST criteria

SECONDARY OUTCOMES:
Objective Response Rate (ORR)_RECIST v1.1 | 24 weeks after the last subject starts CVM-1118
  Assessment by RECIST v1.1 criteria
Duration of response (DoR) | 24 weeks after the last subject starts CVM-1118 up to 1 year after the last-dose
  Duration of response (DoR) is defined as time from the first documentation of response to the time of progression
Progression free survival (PFS) | 24 weeks after the last subject starts CVM-1118 up to 1 year after the last-dose
  Progression free survival (PFS) is defined as time from the first dose of study drug to the time of progression or death
Overall survival (OS) | 24 weeks after the last subject starts CVM-1118 and up to 1 year after the last-dose
  Overall survival (OS) is defined as time from first dose of study drug to death
Time to progression (TTP) | 24 weeks after the last subject starts CVM-1118 up to 1 year after the last-dose
  Time to progression (TTP) is defined as the time from the first dose of study drug to the time of progression
Disease control rate (DCR) | 24 weeks after the last subject starts CVM-1118 and up to 1 year after the last-dose
  Disease control rate (DCR) is defined as the sum of complete response (CR), partial response (PR), and stable disease rate (SD)
Rate of Adverse event (AE) and Serious Adverse Event (SAE) | Starting form the first dose of combination treatment until 28 days (for all AE/SAE) and 90 days (for immune related AE/SAE) following the last dose of treatment by CTCAE v5.
  Rate of Adverse event (AE) and Serious Adverse Event (SAE) are assessed using Common Terminology Criteria for Adverse Events v.5 (CTCAE) criteria
Number of Participants With Abnormal Vital Sign | Starting form the first dose of combination treatment until 28 days (for all AE/SAE) and 90 days (for immune related AE/SAE) following the last dose of treatment
  Values with CTCAE v5 Grade ≧ 3 will be identified with flags. A final outcome result with the number of participants with abnormal vital sign would be provided. Normal ranges will also be provided.
Number of Participants With Abnormal Vital Sign_Assessed the baseline and out-of-range vital signs_ blood pressure (both systolic and diastolic blood pressure) by CTCAE v5 | Starting form the first dose of combination treatment until 28 days (for all AE/SAE) and 90 days (for immune related AE/SAE) following the last dose of treatment
  Both systolic and diastolic blood pressure will be measured. Values with CTCAE v5 Grade ≧ 3 will be identified with flags. A final outcome result with the number of participants with abnormal vital sign would be provided. Normal ranges will also be provided.
Number of Participants With Abnormal Vital Sign_Assessed the baseline and out-of-range vital signs_ Heart rate by CTCAE v5 | Starting form the first dose of combination treatment until 28 days (for all AE/SAE) and 90 days (for immune related AE/SAE) following the last dose of treatment
  Values with CTCAE v5 Grade ≧ 3 will be identified with flags. A final outcome result with the number of participants with abnormal vital sign would be provided. Normal ranges will also be provided.
Number of Participants With Abnormal Vital Sign_Assessed the baseline and out-of-range vital signs_ respiratory rate by CTCAE v5 | Starting form the first dose of combination treatment until 28 days (for all AE/SAE) and 90 days (for immune related AE/SAE) following the last dose of treatment
  Values with CTCAE v5 Grade ≧ 3 will be identified with flags. A final outcome result with the number of participants with abnormal vital sign would be provided. Normal ranges will also be provided.
Number of Participants With Abnormal baseline and out-of range Hematology Count by CTCAE v5 | Starting form the first dose of combination treatment until 28 days (for all AE/SAE) and 90 days (for immune related AE/SAE) following the last dose of treatment
  Values with CTCAE v5 Grade ≧ 3 will be identified with flags. A final outcome result with the number of participants with abnormal laboratory values would be provided. A list of all laboratory normal ranges will also be provided.
Number of Participants With Abnormal Laboratory Values_Assessed the baseline and out-of range coagulation test by CTCAE v5 | Starting form the first dose of combination treatment until 28 days (for all AE/SAE) and 90 days (for immune related AE/SAE) following the last dose of treatment
  Values with CTCAE v5 Grade ≧ 3 will be identified with flags. A final outcome result with the number of participants with abnormal laboratory values would be provided. A list of all laboratory normal ranges will also be provided.
Number of Participants With Abnormal Laboratory Values_Assessed the baseline and out-of range urinalysis test by CTCAE v5 | Starting form the first dose of combination treatment until 28 days (for all AE/SAE) and 90 days (for immune related AE/SAE) following the last dose of treatment
  Values with CTCAE v5 Grade ≧ 3 will be identified with flags. A final outcome result with the number of participants with abnormal laboratory values would be provided. A list of all laboratory normal ranges will also be provided.
Number of patients with abnormalities in electrocardiography (ECG) reporting for PR, QRS, QT, and QTcF intervals | Starting form the first dose of combination treatment until 28 days (for all AE/SAE) and 90 days (for immune related AE/SAE) following the last dose of treatment
  Values with CTCAE v5 Grade ≧ 3 will be identified with flags. A final outcome result with the number of participants with abnormal laboratory values would be provided. A list of all laboratory normal ranges will also be provided.
Maximum Plasma Concentration [Cmax] of CVM-1118 and its metabolite CVM-1125 after CVM-1118 dosing | During Cycle 1 and Cycle 2 (each cycle is 28 days)
  Maximum Plasma Concentration [Cmax] of CVM-1118 and its metabolite CVM-1125 will be measured to see maximum exposure after CVM-1118 dosing
Area Under the Curve [AUC] of CVM-1118 and its metabolite CVM-1125 after CVM-1118 dosing | During Cycle 1 and Cycle 2 (each cycle is 28 days)
  Area Under the Curve [AUC] of CVM-1118 and its metabolite CVM-1125 after CVM-1118 dosing
Pharmacodynamics analysis for the relationship of Cmax and ORR | During Cycle 1 and Cycle 2 (each cycle is 28 days)
  Relationship between Cmax and ORR will be evaluated
Pharmacodynamics analysis for the relationship of AUC and ORR | During Cycle 1 and Cycle 2 (each cycle is 28 days)
  Relationship between AUC and ORR will be evaluated
Pharmacodynamics analysis for the relationship of Cmax and AE | During Cycle 1 and Cycle 2 (each cycle is 28 days)
  Relationship between Cmax and AE will be evaluated
Pharmacodynamics analysis for the relationship of AUC and AE | During Cycle 1 and Cycle 2 (each cycle is 28 days)
  Relationship between AUC and AE will be evaluated

CONTACTS AND LOCATIONS:
Overall Officials: Pei-Jer Chen, MD/PhD, Principal Investigator — National Taiwan University Hospital
Locations (5):
- Taiwan (5):
  - Kaohsiung Chang Gung Memorial Hospital, Kaohsiung City
  - Keelung Chang Gung Memorial Hospital, Keelung
  - National Cheng Kung University Hospital, Tainan
  - National Taiwan University Hospital, Taipei
  - Taipei Veterans General Hospital, Taipei